CLINICAL TRIAL: NCT02872207
Title: Evaluation of the Stinging Potential in Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18196
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suncare agent 1 + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY 987516 (Y65-122); Drug: Control
- Suncare agent 2 + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY 987516 (Y65-118); Drug: Control

INTERVENTIONS:
Drug: BAY 987516 (Y65-122) — 5 µL in one eye
  Arms: Suncare agent 1 + control
Drug: BAY 987516 (Y65-118) — 5 µL in one eye
  Arms: Suncare agent 2 + control
Drug: Control — 5 uL in other eye

SUMMARY:
The objective of this study was to compare the human eye stinging potential of experimental formulas and an industry standard shampoo mixture. The study was conducted under the supervision of a Board Certified Ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 60 years
* No medical conditions of the eyes as determined by the subjects' medical history and confirmed by ophthalmologist
* Subjects do not wear contact lenses or, if he/she does wear contact lenses, is willing to refrain from wearing these during the day of and day after the study
* Subject is willing to have the test materials instilled into the eyes and follow all protocol requirements
* Subject is willing to refrain from using false eyelashes of any type or any topical prescription, OTC or cosmetic products on their eyes, eyelids, eyelashes or the peri-orbital areas of the face on the day of the study.
* Subjects should refrain from use of make-up on testing day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-21 (Actual); Primary Completion 2015-02-22 (Actual); Study Completion 2015-02-22 (Actual)

PRIMARY OUTCOMES:
Subjective discomfort in the eye was assessed based on questions by an Ophthalmologist to the subject, and a 5-category intensity scale. | up to 24 hours
Tearing/Lacrimation was assessed by the Ophthalmologist using a 5-category assessment score for each of the categories | up to 24 hours
Objective inflammation was assessed by the Ophthalmologist using a 5-category assessment score for each of the categories | at 24 hours
Post installation pain/stinging was assessed using a 5-category intensity score | at 24 hours
Post installation itching was assessed using a 5-category intensity score | at 24 hours
Post installation dryness was assessed using a 5-category intensity score | at 24 hours
Post installation scratchiness was assessed using a 5-category intensity score | at 24 hours
Post installation discomfort preventing sleep was assessed using a 5-category intensity score | at 24 hours
Post installation discomfort upon awakening was assessed using a 5-category intensity score | at 24 hours
Post installation excessive discharge upon awakening was assessed using a 5-category intensity score | at 24 hours
Post installation pain in bright sunlight was assessed using a 5-category intensity score | at 24 hours

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerabilitay | at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States